CLINICAL TRIAL: NCT01469208
Title: The Effect of Music Therapy On Infants Born With Gastroschisis
Brief Title: Music Therapy: An Adjunct To Gastroschisis Infants' Care
Acronym: MAGIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Ellen Bendel-Stenzel, Co-Director of NICU research - Minneapolis, Children's Hospitals and Clinics of Minnesota
Other Study IDs: 1110096A
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Gastroschisis
Keywords: Gastroschisis; NICU inpatients; Post surgical repair; Music Therapy
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hope to determine if music therapy will have beneficial effects on physiologic parameters, behavioral states, and pain scale evaluations in infants with gastroschisis defects and if music therapy promotes parental/caregiver relaxation and demonstrates to the parent/caregiver that music is an effective tool to calm and soothe their infant at risk for chronic gastrointestinal discomfort.

Babies will be enrolled during the perinatal period, with therapy to begin after surgical repair of the gastroschisis defect and when the neonatologist deems the baby stable enough for music therapy intervention. Enrolled subjects may receive up to 3 music therapy sessions/week and these sessions may continue until discharge. There is no follow up after discharge.

Each one hour session (20-30 minutes of music and 30 minutes of quiet) will include:

1. Pre music therapy behavior state will be assessed using CRIES scale and recorded.
2. Five minutes of baseline vital signs will be recorded.
3. Music therapy lasting 20-30 minutes, will start. Music therapist will use guitar and lap harp to perform live lullaby tupe music with or with out vocals. Decibel levels will be maintained at 65-75dB. Session will stop if infant shows any signs of distress/agitation. Vital signs will be collected every 1-4 minutes during music session.
4. After session behavior state using CRIES scale will be recorded.
5. Family/caregiver will be given a questionnaire to fill out.
6. 30 min of quiet will start.
7. At the end of quiet time, behavior state and vital signs will be recorded for the last time.

DETAILED DESCRIPTION:
Prior to starting the music therapy session, family/caregivers, if present, will be informed of study session progression. They will be reminded of appropriate behavioral protocol to maintain therapeutic environment during session - i.e. minimal taking & touching, cell phones off etc. A "Do Not Disturb - Music Therapy Session in Progress" will be posted outside pts room on the door.

Behavioral state data and vitals signs collected during sessions will be entered into a database. Also recorded, will be general information about the baby and its mother, such as, gestational age, apgar scores, mothers age and race, number of days post surgical repair etc.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Gastroschisis
2. Patient is stable enough to receive music therapy as determined by Neonatologist
3. Patient has passed their newborn hearing screen

Exclusion Criteria:

1. Neonatologist feels patient/family would not be an acceptable research candidate.

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 30 infants born with gastroschisis will be enrolled over a 2yr period. All babies will be newborns admitted to the NICU. The babies enrolled will be both male and female and diverse in race and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Music Therapy will produce stable physiologic, states as well as, positive behavior states | 3 years
  Vital signs monitor data and stress assessment scores will be collected before, during and post Music Therapy sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospitals and Clinics of MN, Minneapolis, Minnesota, United States